CLINICAL TRIAL: NCT07229391
Title: Examining a Novel Treatment for Persistent Headache After Mild Traumatic Brain Injury
Brief Title: Behavior Therapy vs Education for Persistent Headache After Mild TBI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NURP-008-25S; 1IK2RD001566-01A1 (Other Grant/Funding Number: VA)
Record Dates: First submitted 2025-11-12; First posted 2025-11-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Post-Traumatic Headache
Keywords: Headache; Behavior therapy; Brain Injuries, Traumatic
MeSH Terms: conditions — Post-Traumatic Headache; Headache; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Headache reprocessing (Experimental): Behavior therapy focused on sensations and avoidance behaviors
  Interventions: Behavioral: Headache reprocessing
- Headache education (Active Comparator): Education about ways to limit and manage headaches
  Interventions: Behavioral: Headache education

INTERVENTIONS:
Behavioral: Headache reprocessing — Behavior therapy focused on sensations and avoidance behaviors
  Arms: Headache reprocessing
Behavioral: Headache education — Education about ways to limit and manage headaches
  Arms: Headache education

SUMMARY:
This study will test a new treatment, called Headache reprocessing, for persistent post-traumatic headache. The new treatment will be compared to a headache education intervention. The main objectives of the study are to examine the feasibility, safety, and clinical appropriateness of the new treatment.

DETAILED DESCRIPTION:
Persistent post-traumatic headache (PPTH) is a common, debilitating health condition affecting Veterans and civilians. Relative to other headache disorders, PPTH is especially severe and impairing. PPTH has no established first-line treatments at this time. This research seeks to develop a new behavioral treatment, called headache reprocessing, to target fear and avoidance behaviors and cognitions, and associated neural changes, that drive PPTH. This trial will test the feasibility, safety, and clinical appropriateness of Headache Reprocessing Therapy by comparing it to a headache education control condition in a randomized controlled trial. We will randomize 60 Veterans with PPTH to take part in this study. Headache reprocessing and the educational control intervention will be delivered in group format over eight sessions (one per week for eight weeks). This intervention has the potential to improve available treatment options for PPTH.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in healthcare at VA San Diego Healthcare System;
2. History of mild TBI (mTBI), or head injury that is below the diagnostic threshold for mTBI
3. Headache that had its lifetime onset or significantly worsened within 90 days of a concussive event
4. Headache has persisted for at least 90 days since its onset or worsening
5. No changes in past 3 months to medical management of headache or comorbid psychiatric symptoms, and no anticipated changes during the study interval
6. No current participation in psychological intervention for pain or headache

Exclusion Criteria:

1. History of moderate or severe traumatic brain injury
2. Uncontrolled bipolar, psychotic, or substance use disorder
3. Acute suicidality as determined by screening as "high risk" or has a history of suicide attempt within the past 1 year;
4. Other factors that would preclude participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2027-10-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | Typically up to 3 months, from initial referral to decision to enroll or not
  Number enrolled out of number approached
Attrition | 12 weeks
  % of randomized who are lost to follow-up before week 12
Attendance | During the 8-week intervention
  Percent of participants attending 80+% of sessions
Homework completion | During the 8-week intervention
  Percent of participants completing 80+% of homework
Credibility/Expectancy Questionnaire | Week 12
  Scale measuring how credible the intervention seemed to participants
Client Satisfaction Questionnaire | Week 12
  Scale measuring participant satisfaction with the intervention
Adverse events rated to the intervention | Full study period (28 weeks)
  Adverse events determined to be caused by the intervention
Change in Headache Impact Test-6 score | Week 0 through Week 12
  A widely-used scale measuring the impact that headaches have on daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Fishbein, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Final datasets in machine-readable format will be shared via PubMed Central
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available upon study completion, indefinite
Access Criteria: Public access
URL: https://pmc.ncbi.nlm.nih.gov/